CLINICAL TRIAL: NCT04070716
Title: 3-dimensional Versus 2-dimensional Laparoscopy for Myomectomy: a Randomized Controlled Trial
Brief Title: 3-dimensional Versus 2-dimensional Laparoscopy for Myomectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Taejong Song, Professor, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KBSMC 2019-08-022
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Laparoscopy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D laparoscope (Experimental): For laparoscopic camera system, a 10-mm ENDOEYE FLEX 3D Deflectable Videoscope (Olympus Corp., Germany) was used in the 3D group.
  Interventions: Procedure: 3D laparoscope
- 2D laparoscope (Experimental): For laparoscopic camera system, a 10-mm 30º IDEAL EYES Laparoscope (Stryker, Kalamazoo, MI, USA) camera was used in the 2D group.
  Interventions: Procedure: 2D laparoscope

INTERVENTIONS:
Procedure: 3D laparoscope — For laparoscopic camera system, a 10-mm ENDOEYE FLEX 3D Deflectable Videoscope (Olympus Corp., Germany) was used in the 3D group.
  Arms: 3D laparoscope
Procedure: 2D laparoscope — For laparoscopic camera system, a 10-mm 30º IDEAL EYES Laparoscope (Stryker, Kalamazoo, MI, USA) camera was used in the 2D group.
  Arms: 2D laparoscope

SUMMARY:
The aim of this study is to compare the surgical outcomes and efficacy of 3-dimensional (3D) versus 2-dimensional (2D) imaging systems in laparoscopic myomectomy..

DETAILED DESCRIPTION:
Laparoscopy is founded as a treatment of choice for benign uterine disease. The advantages of laparoscopic surgery over conventional open surgery are less pain, shorter recovery time, shorter hospital stay, and consequently faster return to normal activity as well as better cosmetic effects. However, laparoscopic surgery is more demanding compared with open surgery because operators should project three-dimensional (3D) field through a two-dimensional (2D) monitor.

However, to date, studies examining the possible benefits and drawbacks of 3D imaging system versus 2D in laparoscopic surgery have brought about conflicting results. Moreover, there have been few studies comparing the surgical outcomes of 3D and 2D laparoscopic laparoscopic myomectomy. The aim of this study is to compare the surgical outcomes and efficacy of 3-dimensional (3D) versus 2-dimensional (2D) imaging systems in laparoscopic myomectomy..

ELIGIBILITY:
Inclusion Criteria:

* Uterine myoma requiring laparoscopic myomectomy
* American Society of Anesthesiologists physical status (ASAPS) classification I-II
* absence of pregnancy at the time of surgery.

Exclusion Criteria:

* any suspicious findings of malignant gynecologic diseases,

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2019-08-23 (Actual); Primary Completion 2019-08-23 (Estimated); Study Completion 2019-08-23 (Estimated)

PRIMARY OUTCOMES:
Amount of operative blood loss | At the time of surgery
  Amount of operative blood loss was measured by the anesthesiologists after defining it as the difference between the total amount of suction and irrigation plus the difference between the total gauze weight before and after surgery.

SECONDARY OUTCOMES:
Operative time | At the day of surgery
  Operative time was defined as the time from incision to closure of the skin.

CONTACTS AND LOCATIONS:
Overall Officials: Taejong Song, MD PhD, Principal Investigator — Kangbuk Samsung Hospital, Seoul, Republic of Korea
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No